CLINICAL TRIAL: NCT03467412
Title: A Randomised, Double-blind, Placebo-controlled Phase 2 Trial of FOL-005 to Investigate Efficacy on Hair Growth on Scalp Skin in Healthy Volunteers
Brief Title: To Investigate Efficacy of FOL-005 on Hair Growth on Scalp Skin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Follicum AB (Industry)
Collaborators: Bioskin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FCS-002; 2017-003809-17 (EudraCT Number)
Record Dates: First submitted 2018-03-05; First posted 2018-03-16 (Actual); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-09

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 0.00625 μg FOL-005 (Experimental): 50 μl solution (a total dose of 0.00625 μg FOL-005) injected intradermally three times per week for 12 weeks.
  Interventions: Drug: FOL-005
- 0.025 μg FOL-005 (Experimental): 50 μl solution (a total dose of 0.025 μg FOL-005) injected intradermally three times per week for 12 weeks.
  Interventions: Drug: FOL-005
- 0.050 μg FOL-005 (Experimental): 50 μl solution (a total dose of 0.050 μg FOL-005) injected intradermally three times per week for 12 weeks.
  Interventions: Drug: FOL-005
- 0.100 μg FOL-005 (Experimental): 50 μl solution (a total dose of 0.100 μg FOL-005) injected intradermally three times per week for 12 weeks.
  Interventions: Drug: FOL-005
- Placebo (Placebo Comparator): 50 μl solution (placebo) injected intradermally three times per week for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FOL-005 — intradermal injection
  Arms: 0.00625 μg FOL-005; 0.025 μg FOL-005; 0.050 μg FOL-005; 0.100 μg FOL-005
Drug: Placebo — intradermal injection
  Arms: Placebo

SUMMARY:
The trial was a multicentre, randomised, double-blind, placebo controlled phase 2 trial.

60 healthy bald male subjects diagnosed with alopecia, who are between 18 and 55 years old and provide written informed consent were eligible for inclusion.

The trial period consisted of a screening period of up to 3 weeks followed by 12 weeks of dosing, three times per week. Each subject received two doses of the five trial treatment doses (placebo, 0.00625, 0.025, 0.050, and 0.100 μg respectively). The doses were given as intradermal injections. On each volunteer, two treatment areas were placed on the head and the two selected doses were allocated to the respective treatment areas according to the randomisation scheme. The treatment areas were selected on the border between the bald surface and the surface with hair.

The effect on hair growth was measured by the use of Trichoscan imaging and measuring method at week 8 and 12. A baseline measaure was taken at day 0.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, aged 18-55 years
* Androgenetic alopecia (AGA)) - Norwood/Hamilton grade 3V to 4/4a
* Caucasian, skin type I - IV according to Fitzpatrick's classification

Exclusion Criteria:

* Any dermatological disorders of the scalp which might interfere with the application of Investigational Medical Product or examination method, such as fungal or bacterial infections, seborrheic dermatitis, psoriasis, eczema, folliculitis or scalp atrophy
* Any skin pathology (e.g. scar, nevus) or general condition (e.g. uncontrolled thyroid diseases) that in the investigator's opinion can interfere with the evaluation of the treatment areas or requires topical or systemic therapy
* History of active hair loss due to alopecia areata, scarring alopecia, diffuse telogen effluvium or conditions other than androgenetic alopecia
* Immunological disorders such as alopecia areata, and systemic lupus erythematosus and other systemic known autoimmune disorders
* Diabetes mellitus
* Coagulation deficiencies
* Topical treatments for hair growth (minoxidil, anti-androgens or other agents known to affect hair growth) in the last 6 months
* Topical treatments of the scalp including corticosteroids, tacrolimus, retinoids in the last 2 months or other treatments that may affect hair growth
* Platelet rich plasma (PRP) treatment on scalp during the last 12 months
* Systemic therapy using retinoids, cyclosporine within the last 3 months
* Systemic treatment with beta blockers or corticosteroids, scalp procedures e.g. surgery, laser, light, micro-needling within the last 6 months
* Finasteride (e.g. Propecia®) or Dutasteride intake in the last 12 months, or any systemic hair therapy medication in the last 12 months
* History of any acute (e.g. acute infections) or chronic illness (e.g. psoriasis, atopic dermatitis, porphyria) or known skin cancer that in the opinion of the investigators might confound the results of the trial
* History or clinical signs of keloids or hypertrophic scars
* Positive HIV-Antibody, HBs-Antigen or HCV-Antibody-Test at screening
* Current or within 2 weeks prior to first dosing use of vasodilating drugs (e.g. Pentoxifylline, nitroglycerine) or anticoagulating drugs (e.g. heparins, cumarins, new oral anticoagulants, regular intake of acetylsalicylic acid)
* Current or within 3 months prior to first dosing use of anti-inflammatory medication (ibuprofen, paracetamol is permitted), corticosteroids (nose drops, eye drops and/or inhalers are permitted) or immunosuppressive drugs taken for more than 2 consecutive weeks
* Hair transplantation at any time

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Blume-Peytavi, Professor, Principal Investigator — Klinik für Dermatologie, Charité-Universitätsmedizin, Berlin
Locations (2):
- Germany (2):
  - Klinik für Dermatologie, Venerologie und Allergologie, Charité-Universitätsmedizin, Berlin
  - Bioskin GmbH, Hamburg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each subject received 2 dose strengths on 2 separate areas locally applied on the scalp. Thus, 120 treatment areas were defined in the trial but only 60 subjects participated. The number of participants in each arms are not unique subjects since each subject will appear in 2 arms. The total number of participants in the trial is 60.
Units Other Than Participants: Treatment area on scalp
Period: Overall Study
Arm/Group | 0.00625 μg FOL-005 | 0.025 μg FOL-005 | 0.050 μg FOL-005 | 0.100 μg FOL-005 | Placebo
Started | 25; 25 Treatment area on scalp (Each unique subject will appear in 2 arms. Total sum of subjects is therefore120/2=60.) | 25; 25 Treatment area on scalp (Each unique subject will appear in 2 arms. Total sum of subjects is therefore120/2=60.) | 25; 25 Treatment area on scalp (Each unique subject will appear in 2 arms. Total sum of subjects is therefore120/2=60.) | 25; 25 Treatment area on scalp (Each unique subject will appear in 2 arms. Total sum of subjects is therefore120/2=60.) | 20; 20 Treatment area on scalp (Each unique subject will appear in 2 arms. Total sum of subjects is therefore120/2=60.)
Completed | 22; 22 Treatment area on scalp | 24; 24 Treatment area on scalp | 20; 20 Treatment area on scalp | 23; 23 Treatment area on scalp | 17; 17 Treatment area on scalp
Not Completed | 3; 3 Treatment area on scalp | 1; 1 Treatment area on scalp | 5; 5 Treatment area on scalp | 2; 2 Treatment area on scalp | 3; 3 Treatment area on scalp

BASELINE CHARACTERISTICS:
Population: In total 60 subjects were recruited. However, each subject received 2 treatments which leads up to the total number of subjects appears to be twice as many, i.e. 120.
  Baseline characteristics only reported for the total number of recruited subjects, i.e. 60.
Units Other Than Participants: Areas on the scalp
Groups:
- Combined Baseline Presentation of All Randomised Patient Irrespective of Treatment: In total 60 subjects were recruited. Each subject received 2 treatments in parallell on 2 different treatment areas. Baseline characteristics can therefore not be described for the individual treatment groups as they refer to treatment areas and not subjects. Hence, baseline characteristics are only reported for the total number of recruited subjects, i.e. 60.
Arm/Group | Combined Baseline Presentation of All Randomised Patient Irrespective of Treatment
Number analyzed (Participants) | 60
Number analyzed (Areas on the scalp) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline values were only analysed for the whole study population of 60 subjects
  years | 39.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  Germany | 60
Weight [Mean (Standard Deviation); unit: kg] | 84.91 (14.88)
Height [Mean (Standard Deviation); unit: cm] | 180.6 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Scalp Hair Density
Description: Change from baseline of total hair density (No. of hairs per cm"2") on the scalp
Time Frame: 12 weeks
Population: Note: one subject receiving 0.00625 and 0.050 μg FOL-005 withdrew consent after treatment. Data for primary outcome were available and and consequently used. The nNumber of analysed subjects therefore exceeds number of completed subjects.
Measure: Mean (Standard Deviation); unit: Change from baseline (No. of hairs/cm2)
Arm/Group | 0.00625 μg FOL-005 | 0.025 μg FOL-005 | 0.050 μg FOL-005 | 0.100 μg FOL-005 | Placebo
Number analyzed (Participants) | 23 | 24 | 21 | 23 | 17
Change from baseline (No. of hairs/cm2) | 1.46 (14.75) | 2.58 (15.36) | -4.10 (21.00) | 6.68 (22.24) | 5.60 (16.71)

2. Secondary Outcome: Proportion of Anagen Hairs (%)
Description: Change from baseline in proportion of anagen hairs (%) on the scalp after 12 weeks of treatment. (Only data from subjects included in the PPS are reported.)
Time Frame: From baseline to after 12 weeks treatment
Measure: Mean (Standard Deviation); unit: percentage of anagen hairs
Groups:
- 0.00625 μg FOL-005: 0.00625 μg FOL-005, solution. 50 μl injected intradermally three times per week for 12 weeks.
  FOL-005: intradermal injection
- 0.025 μg FOL-005: 0.025 μg FOL-005, solution. 50 μl injected intradermally three times per week for 12 weeks.
  FOL-005: intradermal injection
- 0.050 μg FOL-005: 0.050 μg FOL-005, solution. 50 μl injected intradermallys three times per week for 12 weeks.
  FOL-005: intradermal injection
- 0.100 μg FOL-005: 0.100 μg FOL-005, solution. 50 μl injected intradermally three times per week for 12 weeks.
  FOL-005: intradermal injection
- Placebo: Placebo. 50 μl injected intradermally three times per week for 12 weeks.
  Placebo: intradermal injection
Arm/Group | 0.00625 μg FOL-005 | 0.025 μg FOL-005 | 0.050 μg FOL-005 | 0.100 μg FOL-005 | Placebo
Number analyzed (Participants) | 23 | 24 | 21 | 23 | 17
percentage of anagen hairs | -0.03 (15.68) | 1.40 (11.43) | -0.73 (14.23) | 3.18 (15.16) | -3.08 (9.53)

3. Secondary Outcome: Change in Proportion of Telogen Hairs (%)
Description: Change from baseline in proportion of telogen hairs (%) on the scalp after 12 weeks of
Time Frame: From baseline to after 12 weeks treatment
Measure: Mean (Standard Deviation); unit: percentage of telogen hairs
Groups:
- 0.050 μg FOL-005: 0.050 μg FOL-005, solution. 50 μl injected intradermally three times per week for 12 weeks.
  FOL-005: intradermal injection
Arm/Group | 0.00625 μg FOL-005 | 0.025 μg FOL-005 | 0.050 μg FOL-005 | 0.100 μg FOL-005 | Placebo
Number analyzed (Participants) | 23 | 24 | 21 | 23 | 17
percentage of telogen hairs | 8.49 (31.36) | -0.05 (22.12) | 8.66 (34.71) | 2.21 (36.82) | 14.60 (25.58)

4. Secondary Outcome: Anagen Hair Density
Description: Change from baseline of anagen hair density (number of hairs per cm"2") on the scalp after 12 weeks of treatment. (Only data from subjects included in the PPS are reported.
Time Frame: From baseline to after 12 weeks treatment
Measure: Mean (Standard Deviation); unit: number of hairs per cm2
Arm/Group | 0.00625 μg FOL-005 | 0.025 μg FOL-005 | 0.050 μg FOL-005 | 0.100 μg FOL-005 | Placebo
Number analyzed (Participants) | 23 | 24 | 21 | 23 | 17
number of hairs per cm2 | -2.26 (28.89) | 3.65 (21.77) | -4.41 (24.85) | 5.79 (25.21) | -2.31 (19.70)

5. Secondary Outcome: Change in Telogen Hair Density
Description: Change from baseline of telogen hair density (number of hairs per cm2) on the scalp after 12 weeks of treatment. (Only data from subjects included in the PPS are reported.)
Time Frame: From baseline to after 12 weeks treatment
Measure: Mean (Standard Deviation); unit: number of hairs per cm2
Arm/Group | 0.00625 μg FOL-005 | 0.025 μg FOL-005 | 0.050 μg FOL-005 | 0.100 μg FOL-005 | Placebo
Number analyzed (Participants) | 23 | 24 | 21 | 23 | 17
number of hairs per cm2 | 3.72 (18.65) | -1.06 (16.33) | 0.31 (16.39) | 0.89 (22.15) | 7.91 (14.34)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Only local adverse events are reported by treatment arm. Systemic adverse events can not be reported by treatment since subjects received two treatments each. These have been reported in a separate group.
Groups:
- 0.00625 μg FOL-005: 0.00625 μg FOL-005, solution. 50 μl injected sub-cutaneous three times per week for 12 weeks.
  FOL-005: intradermal injection
- 0.025 μg FOL-005: 0.025 μg FOL-005, solution. 50 μl injected sub-cutaneous three times per week for 12 weeks.
  FOL-005: intradermal injection
- 0.050 μg FOL-005: 0.050 μg FOL-005, solution. 50 μl injected sub-cutaneous three times per week for 12 weeks.
  FOL-005: intradermal injection
- 0.100 μg FOL-005: 0.100 μg FOL-005, solution. 50 μl injected sub-cutaneous three times per week for 12 weeks.
  FOL-005: intradermal injection
- Placebo: Placebo. 50 μl injected sub-cutaneous three times per week for 12 weeks.
  Placebo: intradermal injection
- Systemic Adverse Events: The systemic (or non-local) AEs are reported for the whole group (60 subjects) only. these events can not be related to one dose strengthe since all subjects received more than one dose.
  Dose range for this group range from 0.0065 μg (subjects receiving a combination of the lowest dose and placebo) to 0.150 μg (subjects receiving a combination of the 2 highest doses)
Arm/Group | 0.00625 μg FOL-005 | 0.025 μg FOL-005 | 0.050 μg FOL-005 | 0.100 μg FOL-005 | Placebo | Systemic Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/20 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/20 | 0/60
Other Adverse Events (participants affected / at risk) | 4/25 | 8/25 | 4/25 | 6/25 | 5/20 | 18/60
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.00625 μg FOL-005 (N=25) | 0.025 μg FOL-005 (N=25) | 0.050 μg FOL-005 (N=25) | 0.100 μg FOL-005 (N=25) | Placebo (N=20) | Systemic Adverse Events (N=60)
Application site eczema (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — General disorders and administration site conditions
Application site exfoliation (General disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) — General disorders and administration site conditions
Application site pustules (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3) | 1 (1) | 4 (5) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (10)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (10)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 5 (5) — General disorders and administration site conditions
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT03467412/Prot_SAP_000.pdf